CLINICAL TRIAL: NCT05536518
Title: Evaluating the Feasibility, Health and Behavioral Impact of Mid-Ohio Farmacy + WW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid-Ohio Food Collective (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20222251
Record Dates: First submitted 2022-08-19; First posted 2022-09-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Food Insecurity; Overweight and Obesity; Produce Prescription; Weight Change, Body
MeSH Terms: conditions — Overweight; Obesity; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mid-Ohio Farmacy (produce prescription) + WW International Coaching (In person and/or Virtual) (Other)
  Interventions: Behavioral: Mid-Ohio Farmacy (produce prescription) + WW International Coaching (In person and/or Virtual)

INTERVENTIONS:
Behavioral: Mid-Ohio Farmacy (produce prescription) + WW International Coaching (In person and/or Virtual) — All study participants are members of the Mid-Ohio Farmacy produce prescription program. All participants are food insecure and will be enrolled and participate in WW coaching sessions for 24 weeks.

SUMMARY:
The aim of this research is to undertake a feasibility study to assess uptake and impact of providing access to a widely available weight management and wellness program (WW; formerly known as Weight Watchers) among individuals experiencing food insecurity and overweight/obesity, who are eligible to receive weekly produce at the Mid-Ohio Food Collective (MOFC) through their pre-existing enrollment in the Mid-Ohio Farmacy program. Participants (n=90) adults over the age of 18 with a BMI between 27-50 kg/m2 will be recruited for a 6 month single-arm clinical trial, where participants will be provided with WW Unlimited Workshop + Digital. The primary objective is to test the feasibility and acceptability of a commercial weight loss and wellness program with an established produce prescription program among individuals experiencing food insecurity and overweight/obesity. Secondary outcomes will include assessments related to weight, height, blood pressure, dietary intake, physical activity, food access, depression, wellbeing and economic factors.

This feasibility study will help inform future interventions among this population. More specifically, this study will help answer questions about the feasibility and acceptability of such an intervention, adherence to the WW program as described to the participant, and the impact that access to a free weight management and wellness program can have on health-related outcomes among individuals experiencing food insecurity and overweight/obesity.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* BMI 27-50 kg/m2
* Positive screen for food insecurity at healthcare provider
* Enrolled in Mid-Ohio Farmacy (produce prescription program)
* Speak English
* Live in greater Columbus,Ohio area for duration of study
* Reliable internet access
* Ability to download and install WW app on phone

Exclusion Criteria:

* Participation in a structured weight loss program in the last 12 months
* WW membership in the last 12 months
* Pregnant, nursing or planning to become pregnant
* Weight loss of 5kg or more in the past 6 months
* Taking prescription medications for weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Total number of patients excluded (Feasibility and Acceptability) | Up to 8 months
  Total number of patients excluded from participation in the intervention
Adherence to study activities (Feasibility and Acceptability) | Up to 8 months
  Percent of study activities completed by each patient
Attrition rate (Feasibility and Acceptability) | Up to 8 months
  Attrition rate (rate at which patients withdraw from the intervention)
Participant Satisfaction with the program (Feasibility and Acceptability) | Up to 8 months
  Participant satisfaction with the intervention (Participant satisfaction questionnaires and semi-structured focus groups)
Food pantry visits (Feasibility and Acceptability) | Up to 8 months
  Total number of food pantry visits prior to and following enrollment in the intervention

SECONDARY OUTCOMES:
Change in body weight (Clinical Outcomes) | Up to 8 months
  Change in body weight (lbs) from the beginning to the end of the intervention
Change in body mass index (BMI) (Clinical Outcomes) | Up to 8 months
  Change in BMI (weight (lb) / [height (in)]2 x 703) from the beginning to the end of the intervention.
Change in blood pressure (Clinical Outcomes) | Up to 8 months
  Change in blood pressure (mmHg) from the beginning to the end of the intervention.
Change in physical activity (Clinical Outcomes) | Up to 8 months
  Change in physical activity (hours/minutes of activity) from the beginning to the end of the intervention.
Change in dietary intake (Clinical Outcomes) | Up to 8 months
  Change in frequency of consumption of fruits/vegetables, whole grain foods and low fat dairy/dairy alternatives from the beginning to the end of the intervention.
Change in food security status (SDOH Outcomes) | Up to 8 months
  Change in food security status from the beginning to the end of the intervention (food secure vs. food insecure)
Change in economic trade-offs (SDOH Outcomes) | Up to 8 months
  Change in economic trade-offs (choices made between purchasing food and other necessities) from the beginning to the end of the intervention
Change in health related quality of life (SDOH Outcomes) | Up to 8 months
  Change in health related quality of life using the CDC Health Related Quality of Life Healthy Days Core Module (HRQOL-4) from the beginning to the end of the intervention
Change in well-being (SDOH Outcomes) | Up to 8 months
  Change in well-being using the World Health Organisation-5 Well Being Index (WHO-5) from the beginning to the end of the intervention.
Change in depression (SDOH Outcomes) | Up to 8 months
  Change in depression using the Patient Health Questionnaire-2 (PHQ-2) from the beginning to the end of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Mid-Ohio Food Collective, Grove City, Ohio, United States

IPD SHARING:
Plan to Share IPD: No